CLINICAL TRIAL: NCT04836650
Title: Effect of Postural Metatarsal Bar Orthotic Element on Stability and Leg Muscular Activity. A Randomized Clinical Trial
Brief Title: Effect of Postural Insoles on Stability and Leg Muscular Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Extremadura (Other)
Responsible Party: Principal Investigator, Alfonso Martínez Nova, Clinical Professor, Universidad de Extremadura
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FOSSIL
Record Dates: First submitted 2021-02-26; First posted 2021-04-08 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Postural Stability; Muscular Activity
Keywords: Metatarsal Bar; Insoles; Postural stability; Electromyograph Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flat Insole (no metatarsal bar) (Placebo Comparator): Postural stability and electromyographic activity in the dominant leg will be assessed with the subject shod (closed clog) and with 1.2 millimeters flat polyester resin insoles.
  Interventions: Diagnostic Test: Postural stability assessment with a force platform.; Diagnostic Test: Muscular assessment with a electromyograph
- Flat Insole (with 2 millimeters metatarsal bar) (Experimental): Postural stability and electromyographic activity in the dominant leg will be assessed with the subject shod (closed clog) and with 1.2 millimeters flat polyester resin insoles with a 2 millimeters polyester resin metatarsal bar.
  Interventions: Diagnostic Test: Postural stability assessment with a force platform.; Diagnostic Test: Muscular assessment with a electromyograph

INTERVENTIONS:
Diagnostic Test: Postural stability assessment with a force platform. — The postural stability will be assessed in static by means of the antero-posterior and medio-lateral displacements of the center of pressure in Romberg open and closed eyes test measured with a force platform (NED/SVE-IBV-Spain). Three 30-second measurements will be made in each condition.
Diagnostic Test: Muscular assessment with a electromyograph — The activity of the medial and lateral gastrocnemius, soleus and anterior tibial muscles of the dominant leg will be assessed with the mDurance surface electromiograph at the same time as postural stability analysis is performed.Three 30-second measurements will be made in each condition.

SUMMARY:
Posturology allows to treat postural problems by using postural insoles, which will have an effect at the neurophysiological level. Pieces of 1 to 3 millimeters are inserted to stimulate specific receptors located on the sole of the foot, which will affect the muscular proprioception and modify the activation of the ascending muscle chains.

The hypothesis of this work is based on the fact that the use of postural insoles with a 2 millimeters metatarsal bar will influence the displacement of the center of pressure and the muscle activity of the leg when compared with a placebo insoles.

Participants will be healthy subjects and will be divided into two groups, control and experimental. Subjects in the control group will be given a pair of flat insoles (placebo insoles) with 1.2 millimeters polyester resin. Those of the experimental group will be made the same insoles but they will include by thermal fusion a metatarsal bar of 2 millimeters polyester resin in the metatarsal zone corresponding to the 1st, 2nd, 3rd and 4th metatarsal head.

Postural stability analysis will be performed with the force platform of the Biomechanics Institute of Valencia (IBV-Spain) and at the same time an electromyographic analysis in the dominant leg with a surface electromyograph system. Subjects will be assessed with their eyes open and closed under two situations, with footwear and with footwear and insoles.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects with no discomfort in gait
* Subjects with not muscle and skeletal diseases

Exclusion Criteria:

* Subjects with balance disorders, pain at legs
* Subjects with loss of balance

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-06 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-22 (Actual)

PRIMARY OUTCOMES:
Change of postural balance | From baseline to 10 minutes
  The mediolateral and anteroposterior excursion of centre of pressures will be measured in millimeters with a force platform with and without the insoles
Change of muscular activity | From baseline to 10 minutes
  The muscular activity in gastrocnemius, soleus and tibialis anterioris will be measured as a percentage (%) with a surface electromyograph in one leg with and without the insoles

CONTACTS AND LOCATIONS:
Locations (1):
- Alfonso Martínez Nova, Plasencia, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No